CLINICAL TRIAL: NCT03939910
Title: The Effect of Preemptive Pudendal Nerve Block Using Bupivacaine Versus Ropivacaine on Post-operative Pain After Posterior Vaginal Repair, Randomized Controlled Trial
Brief Title: Effect of Preemptive Pudendal Nerve Block Using Bupivacaine Versus Ropivacaine on Post-operative Pain After Posterior Vaginal Repair.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Munazzah Rafique (Other Government)
Responsible Party: Sponsor-Investigator, Munazzah Rafique, Physician, King Fahad Medical City
Organization: King Fahad Medical City (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MRafique
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Post-operative Pain After Posterior Vaginal Repair

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): bupivacaine 0.25% for pudendal block
  Interventions: Device: Pudendal Nerve Block needle in pre-packaged kits that include both the trumpet and the needle. The needle will limits its depth of penetration to 5 mm beyond the trumpet.
- Intervention arm (Experimental): ropivacaine 0.2 % for the pudendal block
  Interventions: Device: Pudendal Nerve Block needle in pre-packaged kits that include both the trumpet and the needle. The needle will limits its depth of penetration to 5 mm beyond the trumpet.

INTERVENTIONS:
Device: Pudendal Nerve Block needle in pre-packaged kits that include both the trumpet and the needle. The needle will limits its depth of penetration to 5 mm beyond the trumpet. — Patients will receive a pudendal nerve block injection on each side as previously described 5-10 minutes before the beginning of surgery. A tubular director that allows 1.0-1.5 cm of a 15-cm-long, 22-gauge needle to protrude beyond its tip will be used to guide the needle into the pudendal trunk at lesser sciatic foramen about 1 cm inferior-medial to attachment of the sacrospinous ligament to the ischial spine. The end of the director will be placed against the vaginal epithelium just beneath the tip of the ischial spine. The needle pushed beyond the tip of the director, and 5 ml of the anaesthetic solution will be injected. The needle advanced 1 cm posterior and lateral, and another 5 mL of the anaesthetic solution will be injected into this region.

SUMMARY:
To investigate the efficacy of preemptive pudendal nerve blockade on postoperative pain, after posterior vaginal repair, below the level of ischial spine, excluding uterine suspension procedures that are higher than the coverage of the block.

Primary outcome:

The primary outcome measures of the study visual analogue pain scores and postoperative analgesic consumption.

DETAILED DESCRIPTION:
Preemptive analgesia is widely used during surgical procedures to reduce post-operative pain. Pudendal nerve blockade has been established and provides highly effective and safe anaesthesia to the vulva, lower vagina, and perineum. Various local anaesthetics used in gynaecological practice, including lidocaine, bupivacaine and mepivacaine. Using Bupivacaine in the Pudendal block has shown controversial results. The use of Ropivacaine as preemptive analgesia in different nerve blocks, including nerve block on the face, thorax, abdominal and perineal region, and had shown to be effective.

Bupivacaine and ropivacaine both are commonly used for peripheral nerve blocks. ropivacaine has been shown in two randomized control trials to improved postoperative analgesia and quicker recovery, compared to placebo [28,29]. Previous studies showed the promising effect on different nerve blocks including nerve block on the face, thorax, abdominal and perineal region. However, there are no studies done to investigate the effect of ropivacaine or in comparing their analgesic duration in the setting of a pudendal nerve block for gynaecological surgeries. Therefore, this study aims to conduct a comparison of the duration of postoperative analgesia achieved by two agents.

Therefore, this study aims to conduct a randomized comparison of the duration of postoperative analgesia achieved by pudendal nerve blockade using ropivacaine compared to bupivacaine, in women undergoing posterior vaginal repair. The primary outcome is pain scores and postoperative analgesic consumption, and secondary outcomes include post-operative recovery, ambulation and measure length of hospital stay.

Hypothesis:

Investigators assume that using the Preemptive pudendal nerve block will reduce the postoperative pain and decrease the postoperative analgesic demand in patients who undergo posterior vaginal repair.

The objective:

To investigate the efficacy of preemptive pudendal nerve blockade on postoperative pain, after the posterior vaginal repair, below the level of ischial spine, excluding uterine suspension procedures that are higher than the coverage of the block.

Study Design:

Double-blind randomized controlled trial.

Sample size:

While bearing with the postoperative analgesia consumption (Morphine) over 24 hours as Primary Outcome of interest, presuming Ropivacaine is equivalent to Bupivacaine, the estimated sample size at 95% confidence interval for each arm with 80% power to detect non-inferiority using two-tailed t-test is 30 respectively. Therefore, the total patient required is 60. However, while baring with the 20% patient dropout rate, the estimated sample size for each arm is 36, a total of 72 patients.

Methodology:

Patients will be recruited randomly from urogynecology clinic after fulfilling the inclusion and exclusion criteria, who will undergo posterior vaginal wall repair. Research assistants in the pre-operative anaesthetic clinic will approach patients scheduled for surgery for participation. Patients providing informed consent (Appendix 1) will be allocated to one of two groups using a computer-generated random number table, and blinding of group allocation will be maintained with sequentially numbered, sealed, opaque envelopes. All other personnel - patients, anesthesiologists or caring for the patient in the operating theatre, surgeons, research assistants performing outcome measures, and statisticians - will remain blinded.

The patient will be explained about the risks, benefits and complications and file will be labelled as A or B for that particular patient by computer generated software. The patient can have surgery under spinal or general anaesthesia. Block will be done in the operating room, by the surgeon, just prior to starting the procedure, through the transvaginal approach. One group of patients will receive analgesia, bupivacaine 0.25% to be prepared by the pharmacologist, while the other group will receive ropivacaine 0.2 % in the syringe prepared for the pudendal block. A pharmacist will label syringe as A and B. The enrollment in the study is voluntary.

Work plan:

Pharmacologist role prepare and label two syringes: bupivacaine 0.25% syringe, and Ropivacaine 0.5% syringe. Operating Room nurse will keep two syringes labelled A and B. Before operation nurse will give the surgeon labelled syringe. Postoperatively research nurse will assess the postoperative pain intensity by visual analogue pain scale, as well as analgesic requirements, at 1, 3, 5, 7, 18, 24, and 36 hours.

Pudendal nerve block technique:

All subjects will receive prophylaxis antibiotics [Cefoxitin 2 g intravenously or similar] within one hour before surgery. All surgeries performed transvaginally under general or spinal anaesthesia. Three attending physicians will supervise all surgeries.

Patients will receive a pudendal nerve block injection on each side as previously described 5-10 minutes before the beginning of surgery. A tubular director that allows 1.0-1.5 cm of a 15-cm-long, 22-gauge needle to protrude beyond its tip will be used to guide the needle into the pudendal trunk at lesser sciatic foramen about 1 cm inferior-medial to attachment of the sacrospinous ligament to the ischial spine. The end of the director will be placed against the vaginal epithelium just beneath the tip of the ischial spine. The needle pushed beyond the tip of the director, and 5 ml of the anaesthetic solution will be injected. The needle advanced 1 cm posterior and lateral, and another 5 mL of the anaesthetic solution will be injected into this region. Aspiration will be attempted before every injection to guard against intravascular infusion.

Pain assessment protocols:

investigators will use a validated visual analogue pain scale at 1, 3, 5, 7, 18, 24 and 36 hours after surgery to assess postoperative pain intensity. This pain scale provides a validated and minimally intrusive measure of pain intensity, consisting of a 10-cm vertical line with the two endpoints labelled "no pain" and "worst possible pain." The patient is required to mark the 10-cm line at a point that corresponds to the present level of pain intensity. The distance in centimetres from the low end of the visual analogue scale and the patient's mark are used as a numerical index of pain intensity. To ensure that the questions will be asked in the same way each time, the nursing staff will be trained and instructed to phrase the questions in a standardized fashion, using the specific wording, as follows: "How bad is participant's pain? and mark participant's pain intensity on the pain scale from 0 to 10, where 0 indicates no pain and 10 indicate the worst possible pain. Analgesic requirements will consistently be recorded at 1, 3, 7, 18, and 24 hours after surgery.

Post-operative analgesia:

All patients will be given the following, unless allergic, Paracetamol 1 gm orally every 4 hours, and non-steroidal analgesia in the form of ibuprofen 400 mg orally 8 hourly, to diclofenac 50 mg rectally, 8 hourly, and Tramadol, up to 100 mg orally 8 hourly as required, and analgesia requirement will tabulate in the chart.

Statistical analysis:

Data collection Data will be collected on a customized case report form that includes all relevant demographic and intra-operative data as well as each outcome sought. Patients will be provided with a home diary to complete that will capture all outcomes sought that are not obtained in the hospital. Demographic data will be summarized and expressed using appropriate measures of central tendency and dispersion for continuous data, and frequency for categorical data. The primary outcome, time to the first sensation of pain at the surgical site, will be summarized as mean [SD] or median [IQR] after testing the data for normality with the Kolmogorov Smirnoff test. This will also determine whether groups will be compared with the t-test [for normally distributed data] or Kaplan Meier Survival Curves [for skewed data]. Secondary outcomes that are time-based will also be assessed in the above manner [time to first analgesic request, duration of motor block]. Continuous secondary outcomes [opioid consumption, VRS, room air SpO2] will be assessed with repeated measures ANOVA or the Mann Whitney U-test for non-parametric data. Categorical outcomes will be compared with the Chi-square or Fisher's exact test as necessary.

Ethics:

The approval from the King Fahad Medical City institutional review board [IRB] is taken.

Budget:

Total Budget will be based on estimation according to cost and protocol, and IRF will be obtained

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing posterior vaginal repair.
* Give informed written consent.
* Recruited from the urogynecology department, women specialized hospital, King Fahad Medical City, Riyadh

Exclusion criteria:

* Posterior vaginal repair combined with Uterine suspension procedures [sacrospinous suspension or uterosacral suspension]
* Allergy to high risk to use of bupivacaine or ropivacaine
* coagulopathy
* pre-existing neurologic deficit
* Chronic pain syndromes
* BMI > 40 kg/m2

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing posterior vaginal repair
Enrollment: 72 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
post operative pain assessment | change in pain score from one hour up to 36 hours after surgery will be recorded.
  visual analogue scale for will be used for post operative pain assessment from scale 1 to 10. A higher score indicate worse outcome.
postoperative analgesic consumption. | from one hour up to 36 hours after surgery will be recorded.
  grams or miligrams of intravenous or oral analegesics will be recorded and minimum and maximum amount needed will be recorded. A higher amount indicate worse outcome. An average will be calculated.

SECONDARY OUTCOMES:
Post-operative recovery | up to 6 weeks follow up appointment.
  It will be determined by patient ambulation, return to normal diet and activity and resumption of bowl and bladder function.
Length of hospital stay. | The stay in hospital up to 36 hours to 2 days
  Total number of time spent in hospital
Adverse reaction of analgesic | from 1 hour up to 36 hours postoperatively
  To observe for Potential complications that are rare and include:
  * Hematoma formation from perforation of a blood vessel during needle insertion. Patients with bleeding diatheses may also be at risk.
  * Infection at the site of injection. A localized infection may spread into the retro-psoas space, gluteal muscle, or hip joint
  * Ischial region paresthesia or sacral neuropathy
  * Systemic toxicity after intravascular administration.
Patient satisfaction | up to 6 weeks postoperative followup
  Whether patient is Satisfied, Partially satisfied, Unsatisfied by direct questioning will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided
Need to discuss an ethical committee for feasibility